CLINICAL TRIAL: NCT01952587
Title: Frequency and Functional Impact of the c.32A>T Genetic Polymorphism of TLR7 in Women Infected With HIV-1 : the ANRS EP53 Study
Brief Title: X-linked Biological Response to HIV Sensing: the ANRS EP 53 Study
Acronym: X LIBRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ANRS EP 53 X LIBRIS; 2013-A00954-41 (Other: ANSM (Id RCB))
Record Dates: First submitted 2013-08-05; First posted 2013-09-30 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hiv Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV-infected women (Other): A peripheral blood sample will be collected from HIV-infected women to measure TLR-7 SNP frequency by PCR. IFN-alpha production from pDCs after HIV-1 RNA sensing by TLR7 will also be assessed.
  Interventions: Biological: A peripheral blood sample
- Healthy control women (Other): A peripheral blood sample will be collected from healthy women to measure TLR-7 SNP frequency by PCR. IFN-alpha production from pDCs after HIV-1 RNA sensing by TLR7 will also be assessed
  Interventions: Biological: A peripheral blood sample

INTERVENTIONS:
Biological: A peripheral blood sample — A peripheral blood sample will be collected from HIV-infected subjects and healthy control to measure TLR-7 SNP frequency by PCR. IFN-alpha production from pDCs after HIV-1 RNA sensing by TLR7 will also be assessed

SUMMARY:
Short title :

X-linked biological response to HIV sensing: the ANRS EP 53 study.

Main outcome :

To demonstrate that HIV-infected women carry the TLR7 c.32A>T SNP at a higher frequency than uninfected women, arguing in favor of a role of impaired production of IFN-alpha by pDCs in the risk of becoming infected by HIV-1.

Secondary outcome :

To directly demonstrate at a single cell level that the TLR7 c.32A>T SNP is responsible for a reduce production of IFN-alpha by pDCs after activation of TLR7 by HIV-1 RNA.

Short abstract (public dissemination) :

Male and female display some differences in how their immune system responds to pathogens. This could be related to hormonal or genetic factors located on the X chromosome. This project aims at characterizing X-linked factors that can influence the innate immune response to HIV-1.

DETAILED DESCRIPTION:
Plasmacytoid dendritic cells (pDCs) are key actors of innate immunity that produce high levels of interferon (IFN)-alpha after activation of their Toll-Like Receptors (TLR) by pathogens. A difference between men and women has recently been shown in the level of IFN-alpha produced by pDCs after TLR activation. The production of IFN-alpha in response to TLR7 activation is higher in the presence of estrogens. This could be responsible for gender differences in the level of plasma HIV-1 RNA, that is lower in female as compared to male by about 50%, and for the sex-based differences in the susceptibility to HIV infection. Besides the role of estrogens, X-linked genetic factors could also be involved in the sex-dependent differences in the TLR7-mediated responses of pDCs. TLR7 gene is located on the X chromosome. A single nucleotide polymorphism (SNP) of the TLR7 gene, c.32A>T, have been associated with accelerated disease progression in male HIV patients, and was found over represented in female HIV as well as HCV patients, suggesting that the T allele is associated with a gender-dependent increase of susceptibility to RNA virus infections. A peripheral blood sample will be collected from HIV-infected women and healthy control to measure TLR-7 SNP frequency by PCR. IFN-alpha production from pDCs after HIV-1 RNA sensing by TLR7 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian Female
2. HIV-1 infection (ELISA and western-blot tests)
3. HIV-infection through the sexual route before 50 years-old
4. Continuous antiretroviral therapy for more than 6 months
5. Plasma HIV-1 RNA <50 copies/ml in the last 6 months
6. Age >18-year old
7. Health insurance
8. Informed consent

Exclusion Criteria:

1. HIV-infection through vertical or parenteral routes
2. Chronic infectious disease, notably HCV infection (hepatitis C virus)
3. Acute infectious disease
4. Auto-immune disease
5. Absence of social security (health insurance)
6. Pregnant or breastfeeding woman
7. Incapable adult

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Frequency (%) of subjects carrying the TRL7 c.32A>T SNP in HIV-infected and healthy women | day 1
  arguing in favor of role of impaired production of IFN alpha by pDCs in the risk of becoming infected by HIV 1

SECONDARY OUTCOMES:
Frequency (%) of cells expressing the "A" and "T" alleles of TRL7 in interferon-alpha producing cells | day 1 and month 3

CONTACTS AND LOCATIONS:
Locations (1):
- Purpan Hospital, Toulouse, France

REFERENCES:
- See also: Related Info — http://anrs.fr